CLINICAL TRIAL: NCT06741098
Title: A Study to Evaluate the Safety, Tolerability and Efficacy of NCR100 Injection for the Treatment of Knee Osteoarthritis（ KOA）
Brief Title: A Study of NCR100 Injection for the Treatment of Knee Osteoarthritis（ KOA）
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Collaborators: Shanghai 6th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCR100-1002
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: KOA; Mesenchymal Stromal Cells
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NCR100 injection (Experimental): Subjects will receive four injections of NCR100
  Interventions: Biological: NCR100
- 0.9% Normal saline (Placebo Comparator): Subjects will receive four injections of 0.9% Normal saline
  Interventions: Other: 0.9% Normal saline
- NCR100 injection and 0.9% Normal saline (Experimental): Subjects will receive two injections of 0.9% Normal saline and two injections of NCR100
  Interventions: Biological: NCR100; Other: 0.9% Normal saline

INTERVENTIONS:
Biological: NCR100 — Subjects will receive multiple intra-articular NCR100 injections.
  Arms: NCR100 injection; NCR100 injection and 0.9% Normal saline
Other: 0.9% Normal saline — Subjects will receive multiple intra-articular 0.9% Normal saline injections.
  Arms: 0.9% Normal saline; NCR100 injection and 0.9% Normal saline

SUMMARY:
This clinical study is to investigate the safety and efficacy of NCR100 injection in subjects with knee osteoarthritis (KOA). It contains two parts dose-escalating, and blind random study in adult KOA subjects.

DETAILED DESCRIPTION:
Knee osteoarthritis(KOA) is a kind of degenerative joint disease characterized by chronic inflammation loss of articular cartilage and subchondral bone remodeling.In China, the estimated number of patients diagnosed with KOA reached 37.35millon. The aim of this sudy is to evaluate the safety tolerability and efficacy of human pluripotent stem cell derived mesenchymal stromal cells (NCR100) injection in the treatment of subjects with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and voluntarily sign the Informed Consent Form（ICF） before the enrolment;
* Age: 40-65 years old, both genders;
* Diagnosis of knee osteoarthritis based on American College of Rheumatology criteria;
* Subjects with KOA who have persistent pain for more than six months
* Kellgren-Lawrence grade: II-III

Exclusion Criteria:

* Subjects previously diagnosed of secondary knee osteoarthritis, or those diagnosed with hip/ankle joint disease requiring medical intervention;
* Suffering from other diseases that impair knee function or joints;
* Have received stem cell therapy;
* Have knee injury history;
* Experienced knee surgery, or plan to undergo knee surgery;
* Received analgesics to relieve pain before Investigational Medicinal Product(IMP) injections;
* Have used traditional Chinese medicine to treat KOA within 4 weeks;
* Have used intra-articular injection of drugs to treat KOA within 12 weeks;
* Received glucosamine,chondroitin sulfate, or diacetate therapy before investigational drug intervention within 12 weeks;
* Subjects with acute phase of knee osteoarthritis;
* Severe deformity of the knee;
* Known or suspected allergy or a history of allergies;
* Abnormal results of laboratory examination as follows: Hepatic Insufficiency （Alanine Aminotransferase>2xULN or Aspartate aminotransferase [ast]>2xULN) renal dysfunction (creatinine clearance rate ≤60ml/min or blood urea nitrogen(BUN) > 2× ULN), Coagulation Defects (INR > 1.5) or severe hematological diseases (Grade 3 or above anemia [Hb < 8 g/dL], Grade 2 or above thrombocytopenia platelet count(PLT) < 75×10^9/L) ;
* BMI≥30kg/m^2
* Severe systemic infection or local knee joint infection;
* Have received systemic glucocorticoid therapy before intervention or need to take systemic glucocorticoid therapy during the treatment;
* Have a history of acute myocardial infarction or severe heart diseases,QT prolongation;
* Subjects with peripheral or central nervous system disorders that may interfere assessments;
* Have contraindications to Magnetic Resonance Imaging(MRI)
* Subjects who are unable to walk on his own;
* Subjects with alcohol/drug addiction/abuse or mental disorders;
* Pregnant or lactating, or unable to comply with contraceptives within 6 months after end of study;
* Have participated in other clinical trials within 12 weeks before the screening;
* Severe and poorly controlled comorbidities;

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity(DLT) | 4 weeks after first injection
  Number of participants with Dose-limiting toxicity in 28 days
The Western Ontario and McMaster Universities osteoarthritis index(WOMAC) | 48 weeks after first injection
  Differences of WOMAC scores in changes from baseline between the experimental group and the control group

SECONDARY OUTCOMES:
Adverse Event(AE) or Serious Adverse Event(SAE) | Within 48 weeks of the first infusion
  Number of participants with treatment-related adverse events or serious adverse events assessed by CTCAE v5.0
Visual analogue scale (VAS) | 8 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks
  Differences in changes from baseline between experimental groups and the control group.
Differences in changes from baseline at 8 weeks, 12 weeks, 24 weeks and 36 weeks of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) between the experimental groups and the control group | 8 weeks, 12 weeks, 24 weeks and 36 weeks
  WOMAC scores include three subscale scores (pain, stiffness, and physical function)
Differences in changes from baseline to 24 weeks and 48 weeks in cartilages with various regions | 24 weeks and 48 weeks
  Magnetic resonance imaging (MRI) is used to scan images of knees.